CLINICAL TRIAL: NCT03903835
Title: ProBio: An Outcome-adaptive and Randomized Multi-arm Biomarker Driven Study in Patients With Metastatic Prostate Cancer
Brief Title: ProBio: A Biomarker Driven Study in Patients With Metastatic Prostate Cancer
Acronym: ProBio
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Kom Op Tegen Kanker (Other); Janssen Pharmaceutica N.V., Belgium (Industry); AstraZeneca (Industry); Cancerfonden (Unknown)
Responsible Party: Principal Investigator, Henrik Grönberg, Professor of Cancer Epidemiology, Karolinska Institutet
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT No 2018-002350-78
Record Dates: First submitted 2019-03-29; First posted 2019-04-04 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC); Metastatic Hormone-Sensitive Prostate Cancer (mHSPC)
Keywords: mCRPC; mHSPC; cfDNA; Genomics; Liquid Biopsy
MeSH Terms: interventions — enzalutamide; abiraterone; Abiraterone Acetate; Carboplatin; cabazitaxel; Solutions; Injections; radium Ra 223 dichloride; niraparib; Prednisone; capivasertib; Docetaxel; apalutamide; darolutamide

STUDY DESIGN:
Intervention Model Description: ProBio will use outcome-adaptive randomization, adapting the randomization based on the observed PFS within biomarker signatures. Treatments will initially be assigned to patients based on the biomarker signatures for which that treatment is most likely to be effective. The trial will be analysed within a Bayesian framework, which allows for calculations of the probability for each treatment that is superior to standard of care within a given signature. Each experimental arm will be evaluated for efficacy relative to the control arm with the same biomarker signatures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Control: Standard Care (Active Comparator): Randomization between assignment to the control arm or the biomarker driven arm will be stratified on biomarker signatures, previous treatment, and fraction of ctDNA and will therefore occur after the results from the ctDNA profiling is obtained. Patients in the control arm will receive standard of care following national guidelines.
  Interventions: Drug: Enzalutamide Oral Capsule; Drug: Abiraterone Oral Tablet; Drug: Cabazitaxel 60 mg Solution for Injection; Drug: Docetaxel Injectable Solution; Drug: Radium Chloride Ra-223; Drug: Apalutamide
- Treatment 1 in mHSPC: AR signalling inhibitors (ARSi) (Experimental): Assignments to therapy in the biomarker driven arms will be done on the basis of the biomarker signature using the current information about the efficacy of the various regimens for that signature. Information from previous studies may be incorporated in the randomization at study onset if such reliable data exists. Specifically, patients with an intact androgen receptor (AR) and without TP53 mutations will have increased chance of being randomized to treatment with ARSi.
  Interventions: Drug: Enzalutamide Oral Capsule; Drug: Abiraterone Oral Tablet; Drug: Apalutamide
- Treatment 2 in mHSPC: taxane-based chemotherapy in combination with ARSi (Experimental): Patients with TP53 mutations and TMPRSS2-ERG gene fusions will have an increased chance of being randomised to treatment with chemotherapy plus an ARSi.
  Interventions: Drug: Abiraterone Oral Tablet; Drug: Docetaxel Injectable Solution; Drug: Darolutamide
- Treatment 3 in mHSPC: Poly ADP Ribose Polymerase (PARP) inhibitor (Experimental): DNA-repair deficient patients will have an increased chance of receiving PARP inhibitors at study onset.
  Interventions: Drug: Niraparib plus Abiraterone acetate plus Prednisone
- Treatment 1 in mCRPC: AR signalling inhibitors (ARSi) (Experimental): Specifically, patients with an intact androgen receptor (AR) and without TP53 mutations will have increased chance of being randomized to treatment with ARSi.
  Interventions: Drug: Enzalutamide Oral Capsule; Drug: Abiraterone Oral Tablet
- Treatment 2 in mCRPC: Poly ADP Ribose Polymerase (PARP) inhibitor (Experimental): DNA-repair deficient patients will have an increased chance of receiving PARP inhibitors at study onset.
  Interventions: Drug: Niraparib plus Abiraterone acetate plus Prednisone
- Treatment 3 in mCRPC: selective AKT Inhibitor (Experimental): Patients with alterations in the PI3K pathway will have an increased chance of receiving the combination treatment with Capivasertib plus Docetaxel.
  Interventions: Drug: Capivasertib plus Docetaxel
- Treatment 4 in mCRPC: Carboplatin (Experimental): Only patients with DNA-repair deficiency will be treated with Carboplatin as second line treatment in the castration-resistant phase of ProBio.
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Enzalutamide Oral Capsule — Detailed conditions for the use of the study treatments including dose and dosages are described in accordance with the marketing authorization in the SmPC (Summary of Product Characteristics).
  Other Names: Xtandi
  Arms: Control: Standard Care; Treatment 1 in mCRPC: AR signalling inhibitors (ARSi); Treatment 1 in mHSPC: AR signalling inhibitors (ARSi)
Drug: Abiraterone Oral Tablet — Detailed conditions for the use of the study treatment including dose and dosages are described in accordance with the marketing authorisation in the SmPC.
  Other Names: Zytiga
  Arms: Control: Standard Care; Treatment 1 in mCRPC: AR signalling inhibitors (ARSi); Treatment 1 in mHSPC: AR signalling inhibitors (ARSi); Treatment 2 in mHSPC: taxane-based chemotherapy in combination with ARSi
Drug: Carboplatin — Carboplatin will be administered every 3rd week with an AUC (area under curve) = 5 with a dose calculated according to the Carboplatin AUC Dose calculation (Calvert formula):Dose (mg) = TargetAUC (mg/ml x min) x [GFR ml/min + 25].
  Arms: Treatment 4 in mCRPC: Carboplatin
Drug: Cabazitaxel 60 mg Solution for Injection — Detailed conditions for the use of the study treatment including dose and dosages are described in accordance with the marketing authorisation in the SmPC.
  Arms: Control: Standard Care
Drug: Docetaxel Injectable Solution — Detailed conditions for the use of the study treatment including dose and dosages are described in accordance with the marketing authorisation in the SmPC.
  Arms: Control: Standard Care; Treatment 2 in mHSPC: taxane-based chemotherapy in combination with ARSi
Drug: Radium Chloride Ra-223 — Detailed conditions for the use of the study treatment including dose and dosages are described in accordance with the marketing authorisation in the SmPC.
  Other Names: Xofigo
  Arms: Control: Standard Care
Drug: Niraparib plus Abiraterone acetate plus Prednisone — Niraparib and Abiraterone acetate will be provided by Janssen and will be provided either as a fixed dose combination or as single agents. Detailed use of the study treatment including dose and dosages are described in the Investigator's brochures and SmPC.
  Other Names: Akeega
  Arms: Treatment 2 in mCRPC: Poly ADP Ribose Polymerase (PARP) inhibitor; Treatment 3 in mHSPC: Poly ADP Ribose Polymerase (PARP) inhibitor
Drug: Capivasertib plus Docetaxel — Capivasertib is provided by AstraZeneca and will be given in combination with Docetaxel. All subjects will be given up to ten 21-day docetaxel cycles. All subjects will receive Capivasertib, which will be administered as tablets taken twice a day orally, on a 4 days on/3 days off continuous schedule, commencing cycle one, day 2, until disease progression.
  Arms: Treatment 3 in mCRPC: selective AKT Inhibitor
Drug: Apalutamide — Detailed conditions for the use of the study treatments including dose and dosages are described in accordance with the marketing authorization in the SmPC (Summary of Product Characteristics).
  Other Names: Erleada
  Arms: Control: Standard Care; Treatment 1 in mHSPC: AR signalling inhibitors (ARSi)
Drug: Darolutamide — Detailed conditions for the use of the study treatments including dose and dosages are described in accordance with the marketing authorization in the SmPC (Summary of Product Characteristics).
  Other Names: Nubeqa
  Arms: Treatment 2 in mHSPC: taxane-based chemotherapy in combination with ARSi

SUMMARY:
ProBio is an international, outcome-adaptive, multi-arm, open-label, multiple assignment randomized biomarker driven platform trial in patients with metastatic prostate cancer. Patients will be randomized to control or experimental treatment arms. Patients in the control arm will receive standard of care following national guidelines. Patients in the experimental arm will be randomized to treatments based on a biomarker signature inferred from diagnostic tissue or liquid biopsy profiling. The predefined biomarker signatures are tumor properties or mutations in genes/pathways with previously demonstrated clinical validity (e.g. prognostic value or association with treatment response). The biomarker signatures are identified using a hybridisation capture gene panel specifically designed for prostate cancer.

DETAILED DESCRIPTION:
ProBio is an outcome-adaptive, multi-arm, open-label, multiple assignment randomised biomarker driven platform trial in patients with metastatic hormone-sensitive and castration-resistant prostate cancer.

Patients will be randomised to control or experimental treatment class arms. Patients in the control arm will receive standard of care following national guidelines and will remain within the control arm throughout the course of the trial. Patients in the experimental arm will be randomised to a treatment class (consisting of one or multiple drugs) based on a biomarker signature. The biomarker signatures are defined as tumour properties or mutations in certain genes/pathways identified in the scientific literature as important in prostate cancer treatment response. The biomarker signatures are identified using a gene panel specifically designed for advanced prostate cancer.

Alterations in the following genes/pathways or combinations thereof constitute the biomarker signatures:

* Androgen receptor
* DNA-repair deficiency
* TP53
* TMPRSS2-ERG gene fusion
* PI3K pathway alterations

Patients in the experimental arm can be randomized to the following treatments classes:

for mHSPC

* AR signalling inhibitors (Abiraterone acetate, Enzalutamide, Apalutamide)
* Taxane-based chemotherapy in combination with ARSi (Docetaxel plus Abiraterone acetate, or Darolutamide)
* PolyADP Ribose Polymerase Inhibitors (Niraparib plus Abiraterone Acetate)

for mCRPC

* AR signalling inhibitors (Enzalutamide, Abiraterone acetate)
* Poly ADP Ribose Polymerase Inhibitors (Niraparib plus Abiraterone acetate)
* Selective AKT Inhibitor (Capivasertib plus Docetaxel)

ProBio will use outcome-adaptive randomization, adapting the randomization based on the observed progression free survival (PFS) within biomarker signatures. Treatments will initially be assigned to patients based on the biomarker signatures for which that treatment is most likely to be effective. The trial will be analyzed within a Bayesian framework, which allows for calculations of the probability for each treatment that it is superior to standard of care within a given signature. Each experimental arm will be evaluated for efficacy relative to the control arm with the same biomarker signatures.

Participants and treating physicians will be blinded to ctDNA profile of each patient. The biomarker signatures will thus not influence treatment choice among controls (reflecting today's standard of care).

Further, ProBio will use the sequential multiple assignments trial (SMART) concept, where each patient who progresses within the trial will re-enter the trial and be re-assigned to another treatment based on the patient's current ctDNA profile. Patients will be withdrawn after in total maximal three randomized consecutive treatments after inclusion into the study.

The randomization probabilities within the experimental arm are defined in proportion to the probability that each treatment is superior to standard of care within a given biomarker signature, and therefore change as data accumulates in the trial and knowledge accumulates for what biomarker signatures and specific treatments that are more probable to be effective.

Trial results will be evaluated regularly by an independent data and safety monitoring board (DSMB). The DSMB will evaluate treatment-signature combinations with respect to:

* Graduation for superiority: A treatment-biomarker signature combination will be graduated from the trial if it has a Bayesian predictive probability of success in a future confirmatory phase III trial exceeding a pre-specified threshold (85%).
* Termination for futility: Treatment-biomarker signature combinations will be dropped from the trial for futility when success probabilities drop sufficiently low (less than 10% using a minimum of 20 patients assigned to the specific treatment-biomarker signature combination).
* Alternatively, if the maximum sample size of 300 and 150 patients (for mHSPC and mCRPC, respectively) assigned to a treatment biomarker signature is reached without graduation for superiority, assignments to that combination will end.

ProBio is a platform study. This means that new treatments and biomarker signatures can be added to the experimental arm in the future. This will be done after protocol amendments.

ELIGIBILITY:
Inclusion Criteria:

* Man with histologically confirmed prostate adenocarcinoma, initiating systemic therapy for metastatic disease, encompassing newly diagnosed (i.e. de novo) hormone sensitive prostate cancer (mHSPC) or first-line castration resistant prostate cancer (mCRPC)
* Distant metastatic disease documented by positive bone scan or metastatic lesions on CT or MRI
* Adequate health as assessed by the investigator to receive all available treatments in the trial
* ECOG/WHO (Eastern Cooperative Oncology Group/ World Health Organization) performance score 0-2
* Adequate organ and bone marrow function
* Albumin greater than or equal to 28 g/L
* Able to understand the patient information and sign written informed consent

Exclusion Criteria:

* Other malignancies within 5 years except non-melanoma skin cancer
* Within 6 months of randomization: myocardial infarction, unstable angina, angioplasty, bypass surgery, stroke, TIA (transient ischemic attack), or congestive heart failure NYHA (New York Heart Association) class III or IV
* Uncontrolled hypertension
* Uncontrolled hypotension
* Received systemic therapy (with the exception of standard ADT) prior to study inclusion, for the CRPC indication
* Any severe acute or chronic medical condition that places the patient at increased risk of serious toxicity or interferes with the interpretation of study results
* Unable to comply with study procedures
* Current participation in another clinical trial that will be in conflict with the present study, administration of an investigational therapeutic or invasive surgical procedure within 28 days prior to study enrolment
* Patients who are unlikely to comply with the protocol
* Any condition or situation which, in the opinion of the investigator, would put the subject at risk, may confound study results, or interfere with the subjects participation in this study.
* Any medical condition that would make use of the study treatments contraindicated, according to the SmPC, e.g. significant heart or liver disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) in mCRPC | Until progressive disease or 60 months from start of treatment, whatever occurs first.
  Progression will be evaluated by the established international standards of the Prostate Cancer Working Group version 3 (PCWG3) and for soft tissue metastases (e.g. lung, liver and lymph nodes) according to the Response Evaluation Criteria in Solid Tumors (RECIST v. 1.1).
Progression free survival (PFS) in mHSPC | From date of treatment start until the date of first documentation of progression, assessed up to 60 months
  Time to development of castration-resistance, as defined by EAU guidelines (biochemical progression or radiologic progression)

SECONDARY OUTCOMES:
Treatment response rate in mCRPC | 4 months after treatment start
  Treatment response is evaluated according to PCWG3 and RECIST 1.1
Overall survival (OS) | From enrolment to completion of study (60 months)
  OS is defined as time to death from any cause (overall and prostate cancer specific)
Patient Reported Outcome Measures (PROM) | From enrolment to completion of study (60 months)
  QoL will be assessed using the EORTC QLQ-C30 instrument
Cost-effectiveness | From enrolment to completion of study (60 months)
  Cost effectiveness will be assessed by using the EQ-5D-5L instrument to estimate health utilities. Treatment costs will be based on drug costs and reimbursement data.
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | From enrolment to completion of study (60 months)
  Common Terminology Criteria for Adverse Events (CTCAE) developed and maintained by the US National Cancer Institute will be used to record adverse events
Treatment response rate in mHSPC | 6 months after treatment start
  Response rates at 6 months on therapy will be evaluated by the established standards of EAU Guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Grönberg, Professor, Principal Investigator — Karolinska Institutet; Martin Eklund, Professor, Study Director — Karolinska Institutet; Johan Lindberg, PhD, Study Director — Karolinska Institutet; Piet Ost, Professor, Principal Investigator — University Hospital Ghent, Belgium; Jan Oldenburg, Professor, Principal Investigator — University Hospital, Akershus; Ashkan Mortezavi, MD, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (32):
- Belgium (12):
  - OLV Ziekenhuis Aalst, Aalst
  - GZA Sint-Augustinus, Antwerp
  - AZ Sint-Jan AV, Bruges
  - AZ Sint-Lucas, Bruges
  - Ziekenhuis Oost-Limburg, Genk
  - University Hospital Ghent, Ghent
  - AZ Jan Palfijn Ziekenhuis, Ghent
  - Jessa ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - University Hospital Luik, Liège
  - AZ Damiaan, Ostend
  - VITAZ, Sint-Niklaas
- Norway (5):
  - Ålesund Sjukehus, Ålesund
  - Kreftsenter Kristiansand, Kristiansand
  - Akershus Universitetssykehus, Lørenskog
  - Stavanger Universitetssjukehus, Stavanger
  - Universitetssykehuset Nord-Norge Tromsö, Tromsø
- Sweden (13):
  - Falu lasarett, Falun, Region Dalarna
  - Södra Alvsborgs sjukhus, Borås
  - Länssjukhuset Ryhov - Onkologiska kliniken, Jönköping
  - Länssjukhuset, Kalmar
  - Centralsjukhuset Region Värmland, Karlstad
  - Universitetssjukhuset Örebro, Örebro
  - Karolinska University Hospital, Stockholm
  - Capio St.Görans Hospital, Stockholm
  - Länssjukhuset Sundsvall Härnösand, Sundsvall
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska sjukhuset, Uppsala
  - Hallands sjukhus Varberg, Varberg
  - Centrallasarettet Onkologkliniken, Vaxjo
- Switzerland (2):
  - St. Claraspital, Basel
  - Universitätsspital Basel, Basel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crippa A, Laere B, Discacciati A, Larsson B, Persson M, Johansson S, D'hondt S, Hjalm-Eriksson M, Pettersson L, Enblad G, Ullen A, Lumen N, Karlsson CT, Sandzen J, Janes E, Ghysel C, Olsson M, Sautois B, Schatteman P, Roock W, Bruwaene SV, Verbiene I, Darras J, Everaert E, Maeseneer D, Anden M, Strijbos M, Luyten D, Mortezavi A, Oldenburg J, Ost P, Lindberg J, Gronberg H, Eklund M; ProBio Investigators. Prognostic Value of the Circulating Tumor DNA Fraction in Metastatic Castration-resistant Prostate Cancer: Results from the ProBio Platform Trial. Eur Urol Oncol. 2025 Dec;8(6):1486-1495. doi: 10.1016/j.euo.2025.02.002. Epub 2025 Apr 21. PMID 40263079
- [Derived] De Laere B, Crippa A, Discacciati A, Larsson B, Persson M, Johansson S, D'hondt S, Bergstrom R, Chellappa V, Mayrhofer M, Banijamali M, Kotsalaynen A, Schelstraete C, Vanwelkenhuyzen JP, Hjalm-Eriksson M, Pettersson L, Ullen A, Lumen N, Enblad G, Thellenberg Karlsson C, Janes E, Sandzen J, Schatteman P, Nyre Vigmostad M, Olsson M, Ghysel C, Sautois B, De Roock W, Van Bruwaene S, Anden M, Verbiene I, De Maeseneer D, Everaert E, Darras J, Aksnessether BY, Luyten D, Strijbos M, Mortezavi A, Oldenburg J, Ost P, Eklund M, Gronberg H, Lindberg J. Androgen receptor pathway inhibitors and taxanes in metastatic prostate cancer: an outcome-adaptive randomized platform trial. Nat Med. 2024 Nov;30(11):3291-3302. doi: 10.1038/s41591-024-03204-2. Epub 2024 Aug 20. PMID 39164518
- [Derived] De Laere B, Crippa A, Discacciati A, Larsson B, Oldenburg J, Mortezavi A, Ost P, Eklund M, Lindberg J, Gronberg H; ProBio Investigators. Clinical Trial Protocol for ProBio: An Outcome-adaptive and Randomised Multiarm Biomarker-driven Study in Patients with Metastatic Prostate Cancer. Eur Urol Focus. 2022 Nov;8(6):1617-1621. doi: 10.1016/j.euf.2022.03.005. Epub 2022 Mar 19. PMID 35317973
- [Derived] Crippa A, De Laere B, Discacciati A, Larsson B, Connor JT, Gabriel EE, Thellenberg C, Janes E, Enblad G, Ullen A, Hjalm-Eriksson M, Oldenburg J, Ost P, Lindberg J, Eklund M, Gronberg H. The ProBio trial: molecular biomarkers for advancing personalized treatment decision in patients with metastatic castration-resistant prostate cancer. Trials. 2020 Jun 26;21(1):579. doi: 10.1186/s13063-020-04515-8. PMID 32586393